CLINICAL TRIAL: NCT04977531
Title: H-reflex Measurement in Hemiplegic Stroke Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Heng-Yi, Shen (Other)
Responsible Party: Sponsor-Investigator, Heng-Yi, Shen, Resident of Physical Medicine and Rehabilitation, Cheng-Hsin General Hospital
Organization: Cheng-Hsin General Hospital (Other)
Other Study IDs: (868)110-14
Record Dates: First submitted 2021-07-10; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Stroke; Hemiplegia; Spasticity as Sequela of Stroke
Keywords: H/M slope; H/M maximal amplitude; H/M threshold; stroke; spasticity
MeSH Terms: conditions — Stroke; Hemiplegia; Muscle Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 6 months less: Stroke onset less than 6 months
- 6 months to 2 years: Stroke onset between 6 months and 2 years
- over 2 years: Stroke onset over 2 years

SUMMARY:
As human beings live longer, geriatric disease develop, one of which was stroke whose prevalence elevated by aging. Increased spasticity is a common symptom after stroke and may hinder patient from rehabilitation. The spasticity was evaluated by subjective judgement before. However, in the recent studies, the electrophysiological test, an objective evaluation, showed possibly positive correlation with the spasticity. They compared stroke patients' hemiplegic side with non-hemiplegic side by H/M ratio which showed significant difference. The stroke patients included in studies had stroke onset over 2 years. Therefore, investigators wonder if H/M ratio can evaluate spasticity in stroke patients onset within 2 years and if H/M ratio is correlated to spasticity.

DETAILED DESCRIPTION:
Stroke is a condition that insufficient brain blood supply due to ischemia or hemorrhage causes brain cell death, which impacts normal function of motor, sensory, and speech, depending on the damaged location. Over the world wide, the incidence of stroke is 119 per 100,000 population per year with death rate up to 10-42% in one month after stroke. The survivor developed varying degrees of spasticity up to 42.6%.

In the conventional physical examination, modified Ashworth scale is used to evaluate spasticity, but its results may be influenced by temperature, joints range of motion, subjective judgement by tester or patient's nervousness. In the previous studies, spasticity between hemiplegic side and sound side showed significant difference in ratio of H/M amplitude, H/M threshold and H/M slope. Among them, H/M slope is the most sensitive tool and may be correlated to increased spasticity because H/M slope showed higher value in people with Brunnstrom stage III.

However, patients included in previous studies had disease onset over 2 years. The gold recovery stage after stroke is within 6 months. During this time, many methods can be used to reduce spasticity, such as medicine, stretching exercise, and injection. Therefore, it is very important whether H/M ratio for spasticity evaluation can be performed in patients with disease onset less than 2 years.

In our study, according to onset time, participants will be assigned to three groups: less than 6 months, 6 months to 2 years, and over 2 years. All the participants will accept electrophysiological test over four limbs to collect data of H/M ratio of slope, maximal amplitude and threshold. Hemiplegic side will be compared with sound side for significant difference. The relation between H/M ratio and modified Ashworth Scale will also be identified.

ELIGIBILITY:
Inclusion Criteria:

* Single episode of stroke
* Single side hemiplegia after stroke

Exclusion Criteria:

* Other diagnosis of neurovascular disease or major cardiovascular disease
* Poor cognition
* Poor cooperation
* Aphasia
* People who can not tolerate the exam

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatient or outpatient at department of physical medicine and rehabilitation
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Nerve conduction study (H/M slope) | 30 minutes
  To compare the hemiplegic side and sound side difference, investigators will exam four limbs twice and obtain two data of H and M. Electrodes were placed on each limb and the electrical impulse from low to high ampere will elicit several data of H and M from low to high values. Average of H slope will be calculated and divided by average of M slope, without unit.
Nerve conduction study (H/M maximal amplitude) | 30 minutes
  To compare the hemiplegic side and sound side difference, investigators will exam four limbs twice and obtain two data of H and M. Electrodes were placed on each limb and the electrical impulse from low to high ampere will elicit several data of H and M from low to high values. Maximal H value will be divided by maximal M value, without unit.
Nerve conduction study (H/M threshold) | 30 minutes
  To compare the hemiplegic side and sound side difference, investigators will exam four limbs twice and obtain two data of H and M. Electrodes were placed on each limb and the electrical impulse from low to high ampere will elicit several data of H and M from low to high values. The ampere which elicited first data of H or M will be the threshold. The threshold of H will be divided by the threshold of M, without unit.

SECONDARY OUTCOMES:
H/M slope and modified Ashworth Scale(MAS) | 30 minutes
  Investigators will evaluate if increasing H/M slope is positively correlated with increasing modified Ashworth Scale(MAS). The MAS is used to measure muscle tone, with score of 0, 1, 1+, 2, 3, 4. The higher score means the higher muscle tone.

CONTACTS AND LOCATIONS:
Overall Officials: Szu-fu Chen, MD, PHD, Study Director — Cheng-Hsin General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thrift AG, Thayabaranathan T, Howard G, Howard VJ, Rothwell PM, Feigin VL, Norrving B, Donnan GA, Cadilhac DA. Global stroke statistics. Int J Stroke. 2017 Jan;12(1):13-32. doi: 10.1177/1747493016676285. Epub 2016 Oct 28. PMID 27794138
- [Background] Koton S, Schneider AL, Rosamond WD, Shahar E, Sang Y, Gottesman RF, Coresh J. Stroke incidence and mortality trends in US communities, 1987 to 2011. JAMA. 2014 Jul 16;312(3):259-68. doi: 10.1001/jama.2014.7692. PMID 25027141
- [Background] Bejot Y, Bailly H, Durier J, Giroud M. Epidemiology of stroke in Europe and trends for the 21st century. Presse Med. 2016 Dec;45(12 Pt 2):e391-e398. doi: 10.1016/j.lpm.2016.10.003. Epub 2016 Nov 2. PMID 27816343
- [Background] Hendricks HT, van Limbeek J, Geurts AC, Zwarts MJ. Motor recovery after stroke: a systematic review of the literature. Arch Phys Med Rehabil. 2002 Nov;83(11):1629-37. doi: 10.1053/apmr.2002.35473. PMID 12422337
- [Background] Wissel J, Verrier M, Simpson DM, Charles D, Guinto P, Papapetropoulos S, Sunnerhagen KS. Post-stroke spasticity: predictors of early development and considerations for therapeutic intervention. PM R. 2015 Jan;7(1):60-7. doi: 10.1016/j.pmrj.2014.08.946. Epub 2014 Aug 27. PMID 25171879
- [Background] Stowe AM, Hughes-Zahner L, Stylianou AP, Schindler-Ivens S, Quaney BM. Between-day reliability of upper extremity H-reflexes. J Neurosci Methods. 2008 May 30;170(2):317-23. doi: 10.1016/j.jneumeth.2008.01.031. Epub 2008 Mar 10. PMID 18377996
- [Background] Aloraini SM, Gaverth J, Yeung E, MacKay-Lyons M. Assessment of spasticity after stroke using clinical measures: a systematic review. Disabil Rehabil. 2015;37(25):2313-23. doi: 10.3109/09638288.2015.1014933. Epub 2015 Feb 18. PMID 25690684
- [Result] Funase K, Higashi T, Yoshimura T, Imanaka K, Nishihira Y. Evident difference in the excitability of the motoneuron pool between normal subjects and patients with spasticity assessed by a new method using H-reflex and M-response. Neurosci Lett. 1996 Jan 19;203(2):127-30. doi: 10.1016/0304-3940(95)12284-2. PMID 8834110
- [Result] Walton C, Kalmar J, Cafarelli E. Caffeine increases spinal excitability in humans. Muscle Nerve. 2003 Sep;28(3):359-64. doi: 10.1002/mus.10457. PMID 12929197
- [Result] Phadke CP, Robertson CT, Condliffe EG, Patten C. Upper-extremity H-reflex measurement post-stroke: reliability and inter-limb differences. Clin Neurophysiol. 2012 Aug;123(8):1606-15. doi: 10.1016/j.clinph.2011.12.012. Epub 2012 Jan 23. PMID 22277759
- [Result] Higashi T, Funase K, Kusano K, Tabira T, Harada N, Sakakibara A, Yoshimura T. Motoneuron pool excitability of hemiplegic patients: assessing recovery stages by using H-reflex and M response. Arch Phys Med Rehabil. 2001 Nov;82(11):1604-10. doi: 10.1053/apmr.2001.25081. PMID 11689982